CLINICAL TRIAL: NCT03026244
Title: A Nutritional Intervention Study to Evaluate the Effect of Milk Protein and Prebiotics in Combination With Vitamin D on Innate Immunity in Elderly People
Brief Title: Effect of Milk Protein and Prebiotics in Combination With Vitamin D on Innate Immunity in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL57345.081.16
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-03

CONDITIONS: Immunosenescence; Inflammation
Keywords: Immunity; Elderly; Inflammation; Milk protein; Prebiotics
MeSH Terms: conditions — Inflammation | interventions — Milk Proteins; Prebiotics; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional intervention product (Active Comparator): Milk protein, prebiotics, vitamin D
  Interventions: Dietary Supplement: Milk protein, prebiotics, vitamin D
- Placebo product (Placebo Comparator): placebo product
  Interventions: Dietary Supplement: Placebo product

INTERVENTIONS:
Dietary Supplement: Milk protein, prebiotics, vitamin D — 3 weeks supplementation with milk protein only, followed by 3 weeks milk protein + prebiotics, followed by 3 weeks milk protein + prebiotics + vitamin D
  Arms: Nutritional intervention product
Dietary Supplement: Placebo product — 3 periods of 3 weeks placebo product
  Arms: Placebo product

SUMMARY:
Rationale: The immune system in the ageing population becomes compromised with age (termed "Immunosenescence"). Therefore, elderly people have a decreased ability to respond to infection and vaccination. Furthermore, many of the health issues associated with ageing are linked to inflammation ("Inflammaging"). It has been suggested that this compromised immune function is in part due to reduced Toll-like receptor (TLR) function, which is part of the innate immune system. Milk and dairy based products have been shown to have beneficial effects on inflammation and immunity. This effect may be mediated via support of the innate immune response and promotes TLR7 signaling in in vitro assays (unpublished observation). Also prebiotics have been suggested to influence markers of innate immune function. Furthermore, TLR function has been suggested to be correlated to vitamin D status. Therefore, in the current pilot study, the potential of milk protein, prebiotics and vitamin D to support innate immune function in elderly will be investigated.

Objective: Aim of the current study is to evaluate the effect of milk protein on the innate immune response in elderly in a pilot study. Furthermore, support of this effect by prebiotics and Vitamin D will be studied.

Study design: The study will be a double-blind placebo-controlled pilot study. Study population: Healthy female elderly subjects of 65-85 years of age. Intervention: Period 1: Milk protein or placebo. Period 2: Milk protein + prebiotics or placebo. Period 3: Milk protein + prebiotics + Vitamin D or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 65-85 years
* BMI 20-30 kg/m2
* Non-smoking
* Generally healthy
* Regular and normal Dutch eating habits
* Veins suitable for cannulation (blood sampling)
* Voluntary participation
* Having given written informed consent
* Willing to comply with study procedures
* Accept use of all encoded data, including publication, and the confidential use and storage of all data for 15 years.
* Accept disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Having chronic inflammatory or autoimmune diseases such as rheumatoid arthritis, type 1 diabetes, inflammatory bowel disease
* Disease of GI tract (including major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, known or suspected gastrointestinal disorders, colon or GI tract cancer), liver, gall bladder, kidneys, thyroid gland
* Immune-compromised
* Use of vitamin supplements containing vitamin D and not willing to discontinue this during the study
* Use of anti-inflammatory drugs (for corticosteroids and NSAIDs : frequency >1 per week)
* Use of immunosuppressive drugs
* Excessive alcohol usage (>3 consumptions/day or >15 consumptions/week)
* Participation in any clinical trial including blood sampling and/or administration of substances within 60 days before inclusion in this study
* Use of hormonal replacement therapy
* Mental status that is incompatible with the proper conduct of the study
* A self-reported milk allergy or sensitivity to dairy ingredients
* Unexplained weight loss or weight gain of > 3 kg in the 3 months prior to pre-study screening
* First and second degree relatives of personnel of NIZO food research or Wageningen University, department of Cell Biology and Immunology or Human Nutrition
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results and eventual adverse events to and from his general practitioner
* Holiday to a sunny country during the study, starting from inclusion
* Light therapy during the study, starting from inclusion
* Use of prebiotic supplements during 2 months before study start, and during the study

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Cmax of ex vivo IFN-a production by PBMCs, corrected for baseline | baseline, 3 weeks, 6 weeks, 9 weeks
  Maximum IFN-a levels after 3, 6 and 9 weeks of treatment as compared to baseline in supernatant of PBMCs ex vivo stimulated with TLR ligands.
Cmax of ex vivo IL-6 production by PBMCs, corrected for baseline | baseline, 3 weeks, 6 weeks, 9 weeks
  Maximum IL-6 levels after 3, 6 and 9 weeks of treatment as compared to baseline in supernatant of PBMCs ex vivo stimulated with TLR ligands.

SECONDARY OUTCOMES:
Cmax of ex vivo TNF-a production by PBMCs, corrected for baseline | baseline, 3 weeks, 6 weeks, 9 weeks
  Maximum TNF-a levels after 3, 6 and 9 weeks of treatment as compared to baseline in supernatant of PBMCs ex vivo stimulated with TLR ligands.
Change from baseline in percentage IFN-a producing pDCs | baseline, and highest percentage at either 3 weeks, 6 weeks, or 9 weeks of treatment
  Percentage IFN-a-producing pDCs in PBMCs upon ex vivo stimulation with TLR ligands determined by flow cytometry
Change from baseline in percentage IL-6 producing pDCs | baseline, and highest percentage at either 3 weeks, 6 weeks, or 9 weeks of treatment
  Percentage IL-6-producing pDCs in PBMCs upon ex vivo stimulation with TLR ligands determined by flow cytometry
Change from baseline in percentage TNF-a producing pDCs | baseline, and highest percentage at either 3 weeks, 6 weeks, or 9 weeks of treatment
  Percentage TNF-a-producing pDCs in PBMCs upon ex vivo stimulation with TLR ligands determined by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Els van Hoffen, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO food research, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Splunter M, Perdijk O, Fick-Brinkhof H, Feitsma AL, Floris-Vollenbroek EG, Meijer B, Brugman S, Savelkoul HFJ, van Hoffen E, van Neerven RJJ. Bovine Lactoferrin Enhances TLR7-Mediated Responses in Plasmacytoid Dendritic Cells in Elderly Women: Results From a Nutritional Intervention Study With Bovine Lactoferrin, GOS and Vitamin D. Front Immunol. 2018 Nov 20;9:2677. doi: 10.3389/fimmu.2018.02677. eCollection 2018. PMID 30515164